CLINICAL TRIAL: NCT05977556
Title: The Effect of Perioperative Prehabilitation on Markers of Fitness and Frailty in Patients Undergoing Elective Surgery: a Pilot, Pragmatic, Randomized Controlled Trial
Brief Title: Perioperative Prehabilitation on Markers of Fitness and Frailty in Patients Undergoing Elective Surgery
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: There is another related study that is currently ongoing that would contaminate the control arm.
Sponsor: University of Alberta (Other)
Collaborators: Royal Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00122843
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Neuromuscular strength training: The experimental group will receive up to 24 sessions of neuromuscular strength training led by a physical therapist with expertise in geriatrics and movement behaviors. The program includes exercises such as pelvic lifts, lunges, step-ups, squats, and sit-stands. The difficulty level will progressively increase using techniques like manual resistance, dumbbells, and unstable surfaces.
  Sedentary behavior intervention: The experimental group will also undergo a sedentary behavior intervention based on social cognitive theory. It involves weekly coaching sessions to enhance self-efficacy in reducing sedentary time and increasing light-intensity activity throughout the day. Participants will be provided with a wrist-worn Fitbit activity monitor for daily feedback and to track adherence to the intervention. The aim is to encourage participants to "sit less and move more" throughout their waking hours.
  Interventions: Behavioral: Combined neuromuscular exercise training and 'sit less, move more' program
- Standard of care (No Intervention): The control group will receive standard of care that is provided as part of the perioperative surgical procedure and subsequent rehabilitation.

INTERVENTIONS:
Behavioral: Combined neuromuscular exercise training and 'sit less, move more' program — Neuromuscular strength training: The experimental group will receive up to 24 sessions of neuromuscular strength training led by a physical therapist with expertise in geriatrics and movement behaviors. The program includes exercises such as pelvic lifts, lunges, step-ups, squats, and sit-stands. The difficulty level will progressively increase using techniques like manual resistance, dumbbells, and unstable surfaces.
  Sedentary behavior intervention: The experimental group will also undergo a sedentary behavior intervention based on social cognitive theory. It involves weekly coaching sessions to enhance self-efficacy in reducing sedentary time and increasing light-intensity activity throughout the day. Participants will be provided with a wrist-worn Fitbit activity monitor for daily feedback and to track adherence to the intervention. The aim is to encourage participants to "sit less and move more" throughout their waking hours.
  Arms: Experimental

SUMMARY:
A growing body of evidence suggests that patients who receive good perioperative care (i.e. care prior to surgery, during surgery, and after surgery) tend to have fewer complications, quicker recovery times, and shorter hospital stays. A key component of good perioperative care is recognizing individuals who have diminished physiological reserves (i.e. those who are vulnerable or frail). The stress of an invasive procedure can exhaust the diminished reserves of patients who are frail, which can in turn lead to perioperative complications, mortality and an increase burden to the healthcare system.

Early interventions in patients with diminished reserves can be applied to reduce the risk of complications and poor outcomes. There are emerging studies that show promising benefits of perioperative interventions, such as prehabilitation, though with some mixed findings. Exercise has been shown to reverse or modify the molecular driving factors of frailty, which involve dysregulation of cytokine and endocrine pathways.

Physical inactivity and prolonged sedentary behaviors are also emerging concerns in frailty because of the implicated deleterious health effects. Sedentary behaviors are associated with prevalence and severity of frailty. Among pre-frail and frail inactive adults, sedentary time is associated with higher mortality. Increasing physical activity is recommended as the most feasible approach to prevent and treat frailty. The aim of this study is to determine if a prehabilitation intervention that combines neuromuscular strength training and intervention to reduce sedentary behavior reduces complications, length of stay, and patient recovery, thereby also reducing the burden on the healthcare system.

DETAILED DESCRIPTION:
Frailty is a complex syndrome associated with poor health outcomes in adults, independent of chronological age. Early identification and management of frailty can help improve outcomes and quality of life. Physical activity and exercise interventions, including strength training, have been recommended to manage frailty. Prehabilitation, a preventive intervention before a process of care, has shown promise but with mixed findings. Weight/resistance/strength training and reducing sedentary behavior are important components in frailty management. Sedentary behavior is associated with higher mortality in frail adults. Increasing physical activity may be helpful in preventing and treating frailty. We aim to test a prehabilitation program combining neuromuscular exercise and sedentary behavior intervention in frail adults undergoing elective surgery.

Objective: To evaluate the effect of a 12-week prehabilitation program that combines muscular strengthening exercise with reducing sedentary behaviour for patients 50 years of age or older with frailty undergoing elective surgery.

Hypothesis: The main hypothesis is that the combined prehabilitation program will improve postoperative recovery and reduce the risk of adverse outcomes following elective surgery by improving frailty levels.

Methods: Fifty adults who are vulnerable, mildly, or moderately frail score of 4-6 on the Clinical Frailty Scale (CFS) will be randomly assigned to either the experimental (n=25) or control (n=25) group. The experimental group will receive up to 24 sessions of neuromuscular strength training delivered twice a week over a 12-week period combined with an intervention to reduce and frequently interrupt sedentary behavior. The control group will receive standard of care that is provided as part of the perioperative surgical procedure and subsequent rehabilitation. The "usual care" comparator arm appears to be an appropriate option for a pilot pragmatic study.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* score of 4-6 (vulnerable, mildly or moderately frail) on the clinical frailty scale (CFS)
* scheduled for elective surgery
* ambulatory (indoor and/or outdoor) with or without gait aids

Exclusion Criteria:

* Unstable medical conditions that limit exercise tolerance such as ME/CFS

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline gait speed at 12 and 24 weeks | 12 and 24 weeks
  Comfortable walking speed will be assessed over a 5-meter walkway

SECONDARY OUTCOMES:
Change from baseline physical activity at 12 and 24 weeks | 12 and 24 weeks
  Activpal-derived time spent per day in physical activity
Change from baseline sedentary behavior at 12 and 24 weeks | 12 and 24 weeks
  Activpal-derived time spent per day in sedentary behavior
Change from baseline sleep at 12 and 24 weeks | 12 and 24 weeks
  Activpal-derived time spent per day in sleep
Change from baseline Timed-Up and Go (TUG) test at 12 and 24 weeks | 12 and 24 weeks
  Functional mobility will be assessed using the TUG test
Change from baseline functional lower extremity strength at 12 and 24 weeks | 12 and 24 weeks
  Lower extremity strength will be measured using the 30 seconds sit-stand test
Change from baseline hand grip strength at 12 and 24 weeks | 12 and 24 weeks
  Grip strength will be assessed using a dynamometer
Change from baseline Barthel Index at 12 and 24 weeks | 12 and 24 weeks
  Level of independence in activities of daily living (ADL) will be assessed using Barthel Index
Length of hospital stay after surgery to be determined at 12 and 24 weeks | 12 and 24 weeks
  We will determine the length of stay in the hospital
Readmission rate to hospital after discharge to be determined at 12 and 24 weeks | 12 and 24 weeks
  We will determine the hospital readmissions rate within 30 days of discharge.
Change from baseline Saint Louis University mental status (SLUMS) test | 12 and 24 weeks
  Cognitive assessment will be completed using the SLUMS test
Number of participants with reported postoperative complications | 12 and 24 weeks
  We will determine the number of participants with postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Naheed Rajabali, MD, Principal Investigator — Alberta Health services; Victor Ezeugwu, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No